CLINICAL TRIAL: NCT05774366
Title: Comparative Study of Recovery Characteristics Between Remimazolam Anesthesia With Flumazenil and Desflurane Anesthesia for Closed Reduction of Nasal Bone Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, SO YOUNG LEE, Assistant professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-23-007-L
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — remimazolam; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): receives remimazolam for the maintenance of general anesthesia. At the end of surgery, flumazenil is administered as an antagonist of remimazolam.
  Interventions: Drug: Remimazolam
- Desflurane group (Active Comparator): receives desflurane for the maintenance of general anesthesia.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Remimazolam — General anesthesia was induced with 12 mg/kg/hr of intravenous remimazolam. When loss of consciousness was achieved, the infusion rate of remimazolam was reduced to 1mg/kg/hr for maintenance. At the end of surgery, 0.2 mg of flumazenil is administered.
  Arms: Remimazolam group
Drug: Desflurane — Desflurane (1 minimum alveolar concentration (MAC) of end-tidal desflurane concentration) is used for the maintenance of general anesthesia. Induction of general anesthesia is achieved with 1-2 mg/kg of intravenous propofol bolus.
  Arms: Desflurane group

SUMMARY:
The goal of this prospective, randomized study is to compare recovery characteristics between remimazolam anesthesia with flumazenil and desflurane anesthesia in patients undergoing closed reduction of nasal bone fracture. The main question this study aims to answer is:

* Is there statistically significant difference in time from discontinuation of the anesthetic agent up to patient's response to verbal command between these two groups?

Participants will receive either remimazolam or desflurane for the maintenance of general anesthesia. When the surgery ends, the anesthetic agent will be stopped. For Remimazolam group, flumazenil will be administered as an antagonist of remimazolam.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 75 years
* American Society of Anesthesiologists physical status (ASA PS) of I-II
* Patients undergoing elective closed reduction of nasal bone fracture

Exclusion Criteria:

* Patient who cannot understand the process of this study
* Cognitive, visual or hearing impairment
* Chronic use of antipsychotic medications or medications for sleeping problem
* Use of benzodiazepine
* Patient with kidney or liver disease
* Body mass index (BMI) >30 kg/m^2

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to follow verbal command | from discontinuation of anesthetic agent to response to a verbal command of moving participant's foot, up to 30 minutes
  Time between discontinuation of anesthetic agent and response to a verbal command of moving participant's foot

SECONDARY OUTCOMES:
time to eye opening | from discontinuation of anesthetic agent to eye opening, up to 30 minutes
  Time between discontinuation of anesthetic agent and eye opening
time to extubation | form discontinuation of anesthetic agent to extubation, up to 30 minutes
  Time between discontinuation of anesthetic agent and extubation
Incidence of agitation during emergence period | from discontinuation of anesthetic agent to 2 minutes after extubation
  Ricker Sedation-Agitation Scale (RSAS) >4
Mean arterial blood pressure | from 5 minutes before anesthesia induction to end of anesthesia
  Mean arterial blood pressure measured in the operating room

CONTACTS AND LOCATIONS:
Overall Officials: So Young Lee, M.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea